CLINICAL TRIAL: NCT06941649
Title: Comparison of the Clinical Efficacy of Cervical Single-door Laminoplasty Via the Intermuscular Space Approach and the Conventional Approach: A Multicenter, Prospective Controlled Study
Brief Title: Efficacy of Two Approaches in Cervical Single-door Laminoplasty for Spinal Canal Enlargement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: The First Affiliated Hospital of University of South China (Other); Guangzhou First People's Hospital (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other); The Third Affiliated Hospital of Southern Medical University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYSKY-2025-099-01
Record Dates: First submitted 2025-03-19; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Cervical Spondylotic Myelopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Via the intermuscular space (Experimental)
  Interventions: Procedure: Expansive open-door laminoplasty via intermuscular space approach
- Control (Sham Comparator)
  Interventions: Procedure: cervical single-door laminoplasty via the conventional approach

INTERVENTIONS:
Procedure: Expansive open-door laminoplasty via intermuscular space approach — The cervical laminoplasty via intermuscular space approach will apply bilateral blunt dissection to create the operative space between capital semispinalis muscle and cervical semispinalis muscle
  Arms: Via the intermuscular space
Procedure: cervical single-door laminoplasty via the conventional approach — The cervical laminoplasty via the conventional approach will apply median dissection of the cervical spinous ligament and seperate muscles to expose the whole lamina of cervical vertebrae.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if cervical single-door laminoplasty via the intermuscular space approach can better prevent axial symptom while reaching equal neurological outcome than the conventional approach in adults patients with cervical spondylotic myelopathy. The main questions it aims to answer are:

* Can cervical single-door laminoplasty via the intermuscular space approach better prevent axial symptom than the conventional approach?
* Can cervical single-door laminoplasty via the intermuscular space approach reach the neurological outcome not second to the conventional approach? If there is a comparison group: Researchers will compare the intermuscular space approach and the conventional approach of cervical single-door laminoplasty to see if the intermuscular space approach better prevent axial symptom.

Participants will:

* Received cervical single-door laminoplasty via the intermuscular space approach or the conventional approach once meet the indication.
* Visit the clinic 1 month, 3 months, 6 months, 1 year and 2 years after the surgery.
* Keep a diary of their symptoms and other unexpected conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Patients with cervical spondylotic myelopathy meeting surgery indications.
3. Sign informed consent

Exclusion Criteria:

1. Poor general condition, can not tolerate surgery
2. Patients with long course of disease, degenerative spinal cord, atrophy of limb muscles, and severe joint dysfunction
3. The cervical spine has obvious segmental instability, especially in the case of injury or lesion of the anterior structure, which has not been healed
4. History of cervical spine surgery
5. Combined with obvious cervical kyphosis
6. Combined with cervical fracture, dislocation, etc
7. Combined with cervical spinal infection, arthritis and other pathological changes
8. Combined with tumors of cervical spine or spinal cord.
9. Mental retardation or other causes of limited behavioral ability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
modified Japanese Orthopedic Association score | 2 years after operation
  Evaluate neurological function in 4 dimension with a total of 18 points:
  A. Upper limb motor dysfunction(5 points) B. Lower limb motor dysfunction(7 points) C. Sensory dysfunction(3 points) D. Sphincter dysfunction(3 points)

SECONDARY OUTCOMES:
modified Japanese Orthopedic Association Score | Before surgery and 1week, 1month, 3months, 6months, 1year after surgery
  Evaluate neurological function in 4 dimension with a total of 18 points:
  A. Upper limb motor dysfunction(5 points) B. Lower limb motor dysfunction(7 points) C. Sensory dysfunction(3 points) D. Sphincter dysfunction(3 points)
Cervical Visual Analogue Scale Score | Before surgery; 1week, 1month, 3months, 6months, 1year and 2 years after surgery
  According to the severity of patient's neck pain, on a scale of 1-10, let patients themselves choose one score.
  0 means no pain and 10 means extreme pain.
Zeng's axial symptom scale | Before surgery; 1week, 1month, 3months, 6months, 1year and 2 years after surgery
  Based on the impact on work and life, and objective examination of neck paraspinal muscles and trapezius for spasms and tenderness, divided into 4 grades:
  * "Excellent": No abnormal sensations in the neck, no tenderness or muscle spasms;
  * "Good": Mild symptoms after fatigue or cold exposure, but quick recovery, no significant impact on daily work and life, no tenderness or mild spasms in neck muscles, no need for painkillers;
  * "Fair": Symptoms often appear <100 days/year, daily work and life are somewhat affected, mild tenderness or spasms in neck muscles, need for painkillers with good effect;
  * "Poor": Symptoms frequent (>100 days/year), significantly affecting daily work and life, obvious tenderness or spasms in neck muscles, need for painkillers with poor effect.
  Those rated as excellent and good are considered to have no axial symptoms, while those rated as fair and poor are considered to have axial symptoms, and the incidence is calculated.
Hosono axial symptom scale | Before surgery; 1week, 1month, 3months, 6months, 1year and 2 years after surgery
  According to patients' axial symptom and which treatment can alleviate it:
  Severe (regular need for analgesics or local injections), Moderate (regular need for physical therapy or compression), or Mild (no need for treatment). Severe and moderate are defined as having axial symptoms, while mild is defined as having no axial symptoms.
Cervical 11-point Numerical Rating Scale | Before surgery; 1week, 1month, 3months, 6months, 1year and 2 years after surgery
  Based on neck symptoms, ask the patient to rate their condition on a scale from 0 to 10, where 0 indicates no symptoms and 10 indicates severe symptoms

OTHER OUTCOMES:
Incidence of adverse reactions | 1 week, 1month, 3months, 6months, 1year and 2 years after surgery
  Safety Metrics Incidence of adverse reactions= (amount of adverse reactions/amount of patients)*100%
Incidence of adverse events | 1 week, 1month, 3months, 6months, 1year and 2 years after surgery
  Safety Metrics Incidence of adverse events= (amount of adverse events/amount of patients)*100%
Incidence of severe adverse events | 1 week, 1month, 3months, 6months, 1year and 2 years after surgery
  Safety Metrics Incidence of severe adverse events= (amount of severe adverse events/amount of patients)*100%
Mortality | 1 week, 1month, 3months, 6months, 1year and 2 years after surgery
  Safety Metrics Mortality= (amount of death/amount of patients)*100%